CLINICAL TRIAL: NCT05612841
Title: A Study on Drug-drug Interactions in Patients Treated With Anticancer Agents for a Non Metastatic Castrate-resistant Prostate Cancer or a Metastatic Castrate naïve Prostate Cancer in Real Life Setting
Brief Title: A Study on Drug-drug Interactions in Patients Treated With Anticancer Agents for a Prostate Cancer in Real Life Setting
Acronym: IN-PROVE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/660
Record Dates: First submitted 2022-02-23; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Prostatic Neoplasm
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- non metastatic castration resistant prostate cancer
  Interventions: Other: data collection
- metastatic castrare naïve prostate cancer
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — data collection from drug-drug interaction between anti-cancer treatment and and other medications

SUMMARY:
This will be a national observational, non-randomised, multicentre study, conducted in France.

Patients will be recruited in routine clinical practice by office- or hospital-based urology and/or oncology specialists when a first line treatment for their castrate resistant prostate cancer is initiated. The decision to treat patients with either agent preceding study enrolment will be left to the investigator's decision, per routine clinical practice. The nature of treatment and clinical care of patients will not be influenced by their participation in the study. All patients meeting the study criteria who visit the study physician will be consecutively invited to participate in the study to minimise recruitment bias. All medications administered will be collected. This is a non-interventional study. The investigators are free to choose products, and modalities of administration in accordance with the local Summary of Product Characteristics Therefore, the decision to prescribe one of these therapies must be made prior to and independently from the decision to enrol patients in this non interventional study.

Potential DDI will be identified using electronic screening methods (Micromedex Software and Theriaque Software).

This design will enable assessment of treatment and subsequent outcomes based on local standards, and is likely to encompass a wider range of therapeutic decisions compared with the stricter, defined limits on therapy required by investigational study protocols. Decisions and outcomes made in real-world conditions are likely to be more widely applicable to clinical practice than those from interventional studies.

Following French regulation there is no need for an approval of ethic committee for this type of observational study.

ELIGIBILITY:
* Males aged ≥18 years;
* Histologically or cytologically confirmed diagnosis of adenocarcinoma of the prostate
* For patients with a nmCRPC, documented castration resistance with progression of prostate cancer on androgen deprivation therapy (ADT) (surgical or chemical);
* Initiation of first- line systemic therapy (with abiraterone, apalutamide, darolutamide, docetaxel or enzalutamide) for a non metastatic castrate-resistant or a metastatic castrate naïve prostate cancer according to the approved labels and current guidelines. The metastatic status is based on conventional imaging (CT scan, bone scan).

Patients are not eligible if they are receiving an investigational treatment for prostate cancer of any kind.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a non metastatic castration-resistant or a metastatic castrate naïve prostate cancer, with a minimum of 100 patients with a non metastatic castrate-resistant prostate cancer.
Sampling Method: Probability Sample
Enrollment: 264 (Estimated)
Dates: Start 2022-04-05 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with a non metastatic castration-resistant or a metastatic castrate naïve prostate cancer with at least one significant drug interaction. | 18 months

SECONDARY OUTCOMES:
Total number of drug interactions per patient | 18 months
  Hatoum scale: level 1 to level 4
Description of the rate of patients with prostate cancer presenting a significant comorbidity according to investigator in a real life setting | 18 months
Exploratory assessment of baseline clinical (e.g. age, comorbidities, stage of cancer, ECOG) or biological (e.g. CBC, liver tests, PSA, albumin) parameters that may be link to a higher risk of drug interaction | 18 months
  assessed either by the Micromedex software or the national thesaurus of the ANSM

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No